CLINICAL TRIAL: NCT07052162
Title: Safety, Pharmacokinetics, and Preliminary Efficacy of Tafenoquine for the Treatment of Vivax Malaria in Papua New Guinean Children
Brief Title: Investigating the Pharmacokinetics of Tafenoquine in Healthy Papua New Guinean Children
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES67418
Record Dates: First submitted 2025-03-27; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Pharmacokinetics of Tafenoquine
Keywords: tafenoquine; vivax malaria; pharmacokinetics; children
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Water; CD36 Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Single-dose tafenoquine as 10 mg/kg taken with water and a low-fat meal (3 plain cracker biscuits; 2% fat)
  Interventions: Drug: Single dose tafenoquine (10 mg/kg) given with water
- Group B (Experimental): Single-dose tafenoquine as 10mg/kg taken with 250 mL chocolate flavoured milk (9% fat) and a low-fat meal (3 plain cracker biscuits; 2% fat).
  Interventions: Drug: Single dose tafenoquine (10 mg/kg) given with fat

INTERVENTIONS:
Drug: Single dose tafenoquine (10 mg/kg) given with water — Participants will receive single-dose TQ as 10 mg/kg taken with water and a low-fat meal (3 plain cracker biscuits; 2% fat). Food (low-fat meal) is taken with both regimens to attenuate any gastrointestinal adverse effects that are related to taking TQ on an empty stomach. Combinations of full or half-tablets will be swallowed whole or crushed lightly (tablets) or dissolved in boiled water (if dispersible tablets are available), as directly observed treatment. Children vomiting within the first 30 minutes of treatment will be withdrawn
  Other Names: TQ; Tafenoquine succinate; Kodatef
  Arms: Group A
Drug: Single dose tafenoquine (10 mg/kg) given with fat — Single-dose TQ as 10 mg/kg taken with 250 mL chocolate flavoured milk (9% fat) and a low-fat meal (3 plain cracker biscuits). Food (low-fat meal) is taken with both regimens to attenuate any gastrointestinal adverse effects that are related to taking TQ on an empty stomach. Combinations of full or half-tablets will be swallowed whole or crushed lightly (tablets) or dissolved in boiled water (if dispersible tablets are available), as directly observed treatment. Children vomiting within the first 30 minutes of treatment will be withdrawn
  Other Names: TQ; Tafenoquine succinate; Kodatef
  Arms: Group B

SUMMARY:
Plasmodium vivax is the most geographically widespread malaria species and the second largest contributor to symptomatic malaria worldwide. It accounts for half of all malaria cases outside Africa, with an estimated 14.3 million clinical vivax malaria cases reported annually, contributing to an annual cost of US$359 million. Children are most vulnerable to infection, with P. vivax prevalence peaking between 2 to 6 years of age. In Papua New Guinea (PNG), there are >1.5 million suspected P. vivax cases annually, and while P. falciparum infections are the most prevalent, P. vivax transmission is the most intense in the world. P. vivax in PNG provides a unique epidemiological setting in which to assess innovative treatments in children.

The complex biology of P. vivax represents a challenge for malaria control and chemotherapy, especially dormant liver-stage parasites (hypnozoites) which can reactivate (relapse) and cause disease at a time remote from the primary infection. Hypnozoite relapse is the primary cause of vivax malaria in endemic regions and is resistant to most antimalarial drugs. Identifying effective treatments for radical cure, the complete elimination of parasites (both blood- and liver-stage), is therefore a priority. The World Health Organization (WHO) recommends a 14-day radical cure regimen for uncomplicated vivax malaria; comprised of blood stage treatment (chloroquine or artemisinin combination therapy (ACT)) and 14 days of the 8-aminoquinoline drug primaquine (PQ; 0.25-0.5 mg/kg/day) for liver-stage cure. More recently, the 8-aminoquinoline tafenoquine has garnered interest as an alternative radical cure agent to primaquine. However, there is limited data on the pharmacokinetics, tolerability and radical cure efficacy of tafenoquine in children.

The overall aim of the study is to characterise the pharmacokinetic profile of tafenoquine (and primary metabolite) in Papua New Guinean children.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the pharmacokinetic disposition of tafenoquine, with and without coadministration of fat, in healthy Papua New Guinean children. This study represents the first part of a multi-phase evaluation of tafenoquine in PNG children (preliminary efficacy study registered separately).

In this study, healthy PNG children aged 5-12 year will be eligible for inclusion into the study providing they have normal G6PD activity (>70% enzyme activity) and no history of previous hypersensitivity to 8-aminoquinoline drugs. All participants will be admitted to the Alexishafen Health Centre for the first 2-4 days of the study, to facilitate blood sampling and clinical monitoring.

After admission, baseline demographic and medical history will be taken, and the participants will undergo a full clinical assessment to establish baseline safety indices. The 30 participants will then be randomized 1:1 to receive either:

Group A: single dose tafenoquine (10 mg/kg) with water (and cracker biscuits (2% fat), to mitigate gastrointestinal complaints, or Group B: single dose tafenoquine (10 mg/kg) with 250mL of chocolate flavoured mild (9% fat; and cracker biscuits (2% fat)).

For pharmacokinetic analysis, venous blood samples will be collected (via indwelling cannula) at 8 time points within the first 48-hours of drug administration, with further finger prick samples collected on days 3, 4, 7, 14, 28, 42 and 56. Both dried blood spot and plasma samples will be collected at all time points for pharmacokinetic analyses.

Standardised review, including adverse-effect questionnaires, and clinical monitoring (haemoglobin, methaemoglobin, reticulocyte counts, malaria blood films) will be conducted at all daily follow-up time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, and 56). Safety testing (hepatorenal function tests (ALT, total bilirubin, creatinine), haemoglobin, urine dipstick analysis and electrocardiogram trace, will be taken at 4, 12, 24 hours and on Days 3, 7 and 28. A standardized clinical taste evaluation survey will be conducted (child or parent response, age dependent) 30 minutes of dosing, which will be repeated on Day 1.

Secondary objectives:

1. To evaluate the role of fat on the bioavailability of tafenoquine
2. To assess the safety of tafenoquine in PNG children
3. To assess the tolerability of tafenoquine in PNG children

The investigators hypothesise that:

1. A single dose of tafenoquine (10 mg/kg) is safe in PNG children
2. Co-administration of tafenoquine with fat will improve drug bioavailability
3. Cut or crushed tablets will not be well tolerated, although tolerability will improve with administration of whole tablets

ELIGIBILITY:
Inclusion Criteria:

* have a normal glucose-6-phosphate-dehydrogenase (G6PD) activity (>70% enzyme activity) as confirmed by quantitative SD Biosensor
* are Rapid Diagnostic Test negative for malaria
* have not received treatment with any antimalarial in the previous 4-weeks
* have no signs or symptoms of significant morbidity
* have no history of hypersensitivity to primaquine
* are able to attend all scheduled follow-up visits

Exclusion Criteria:

* have G6PD activity <70%
* test positive for malaria by rapid diagnostic test
* have receive treatment with an antimalarial in the previous 4-weeks
* have signs or symptoms of significant morbidities
* have a history of primaquine related hypersensitivity
* cannot, or are not willing, to attend all scheduled follow-up visits

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: Distribution half-life | 56-days after drug administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from venous blood samples collected at baseline (Day 0), 2, 4, 8, 12, 18, 24, 36 and 48 hours from a sampling cannula with capillary finger-prick samples at Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetic: Terminal elimination half-life | 56-days after drug administration
Pharmacokinetic: Absorption half-life | 56-days after drug administration
Pharmacokinetics: Clearance | 56-days after drug administration
Pharmacokinetics: Volume of distribution | 56-days after drug administration
Pharmacokinetics: Maximal concentration | 56-days after drug administration
Pharmacokinetics: Area under concentration-time curve | 56-days after drug administration

SECONDARY OUTCOMES:
Safety: Change in haemoglobin over 28 days | 28-days from drug administration
  After admission, baseline demographic details (age, weight, height) and a detailed clinical history will be taken. All participants will then undergo a full clinical assessment, documenting axillary temperature, heart and respiration rate, and methaemoglobin level (pulse oximetry; Rad57 pulse oximeter with SpMet% function). A blood sample will be drawn prior to drug administration via the cannula for baseline laboratory tests (safety analysis) and genotyping, including:
  i) Haemoglobin and blood glucose ii) Dipstick urinalysis iii) Resting 12-lead electrocardiogram for rate-corrected QT interval iv) 250 μL blood sample for CYP2D6 genotyping v) Reticulocyte count vi) Hepatorenal function Safety testing, including collection of a 100 μL blood sample for hepatorenal function tests (ALT, total bilirubin and creatinine), haemoglobin, methaemoglobin, urine dipstick analysis (blood, protein and glucose), and an electrocardiogram trace, will be taken at 4, 12, 24 hrs, and on Days 3, 7 and 28.
Safety: Change in methaemoglobin over 28 days | 28-days from drug administration
Safety: Change in hepatorenal function over 7 days | 7-days from drug administration
Safety: Change in rate corrected QTc over 28 days | 28-days from drug administration
Tolerability: Taste and tolerability assessment | 1-day following drug administration
  A standardized clinical taste evaluation/tolerability survey will be conducted (child or parent response, dependent on age) 30 minutes after TQ dosing, which will be repeated on Day 1. This survey will investigate the participant's feelings towards the dosing experience (taste, tablet size, ease of swallowing) and any treatment related side effects (focussing on known complications including nausea, gastrointestinal disruption, vomiting).
Safety and tolerability: Number of participants with treatment-related adverse events as assessed by standardised questionnaire | 56-days after drug administration
  Symptom questionnaires (used across all research conducted at this site) will be conducted at each follow-up time point from baseline (Day-0) until end of study (day 56). The questionnaire will determine the frequency, duration and rating (mild, moderate, severe) of each adverse event experienced, from the perspective of the participant/caregiver and clinic staff.

CONTACTS AND LOCATIONS:
Overall Officials: Brioni R Moore, PhD, Principal Investigator — Curtin University
Locations (1):
- Alexishafen Health Centre, Madang, Madang Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: No
Data maybe shared upon contact with the principal investigators and approval by the PNG Institute of Medical Research. This process will be conducted on a case by case basis, as per agreements between collaborative partners.